CLINICAL TRIAL: NCT06477198
Title: Posterior Quadratus Lumborum Block vs Erector Spinae Plane Plane Block for Pain Management After Lumbar Spinal Surgery
Brief Title: QLB vs ESPB for Lumbar Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 37
Record Dates: First submitted 2024-06-13; First posted 2024-06-27 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar Disc Herniation; Postoperative pain management; Erector spinae plane block; Quadratus lumborum block
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: Sixty patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification I-II and scheduled for lumbar disc herniation surgery will be included in the study. Patients will be randomly divided into two groups (Group QLB = QLB group, Group ESPB = ESPB group) including 30 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes Assessor and participant were blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group QLB = QLB group (Active Comparator): Posterior QLB will be performed
  Interventions: Other: QLB; Other: Postoperative analgesia management
- Group ESPB = ESPB Group (Active Comparator): Lumbar ESPB will be performed
  Interventions: Other: ESPB; Other: Postoperative analgesia management

INTERVENTIONS:
Other: QLB — The block procedure will be applied after the surgery and before extubation with patients in the prone position by using US (Vivid Q, GE Healthcare, US). Under aseptic conditions, the convex probe will be covered with a sterile sheath and a 22G, 80 mm block needle (Braun Stimuplex Ultra 360, Germany) will be used. After visualizing the quadratus lumborum muscle, the needle will be punctured and 5 ml of saline will be injected into the posterior border of the quadratus lumborum muscle between QLM and latissimus dorsi muscle.. After the block location is confirmed, 30 ml of 0.25% bupivacaine will be injected. The same process will be applied to the opposite side (60 ml totally).
  Arms: Group QLB = QLB group
Other: ESPB — ESP block will be performed. Convex probe will be placed longitudinally 4 cm lateral to the L3 transverse process. Erector spinae muscle will be visualized on the hyperechoic transverse process. The block needle will be inserted cranio caudal direction and then for correction of the needle, 2 ml saline will be injected deep into the erector spina muscle fascia. Following confirmation of the correct position of the needle 30 ml %0.25 bupivacaine will be administered for the block in each side (total 60 mL).
  Arms: Group ESPB = ESPB Group
Other: Postoperative analgesia management — Patients will be administered paracetamol 1 gr IV every 8 hours in the postoperative period. Postoperative patient evaluation will be performed by a pain nurse blinded to the procedure. Tramodol will be performed for rescue analgesia.

SUMMARY:
Ultrasound-guided quadratus lumborum block (QLB) is a fascial plane block where local anesthetic is injected adjacent to the quadratus lumborum muscle to anesthetize the thoracolumbar nerves.

The ultrasound (US) guided erector spina plane block (ESPB) is a novel interfacial plan block defined by Forero et al. at 2016. Visualization of sonoanatomy with US is easy, and the spread of local anesthesic agents can be easily seen under the erector spinae muscle. Thus, analgesia occurs in several dermatomes with cephalad-caudad way. It has been reported that ESPB provides lumbar analgesia at T10-12, L3.

This study aims to compare US-guided ESPB and posterior QLB for postoperative analgesia management after lumbar disc herniation-laminectomy surgery.

DETAILED DESCRIPTION:
Spine surgery in thoracolumbar region is one of the most common surgeries performed for the treatment of leg and back pain. Pain management is especially important for these patients since chronic pain often occurs after surgery. Severe pain may occur at postoperative period in patients following lumbar disc herniation (LDH) operation. Postoperative effective pain treatment provides early mobilization and shorter hospital stay, thus complications due to hospitalization such as infection and thromboembolism may be reduced.

Opioids are one of the most preferred drugs among the analgesic agents. Parenteral opioids are generally performed for patients after surgery. However opioids have undesirable adverse events such as nausea, vomiting, itching, sedation and respiratory depression (opioid-related adverse events).

Various methods may be performed to reduce the use of systemic opioids and for effective pain treatment. US-guided interfascial plane blocks have been used increasily due to the advantages of ultrasound in anesthesia practice. Ultrasound-guided quadratus lumborum block (QLB) is a fascial plane block where local anesthetic is injected adjacent to the quadratus lumborum muscle to anesthetize the thoracolumbar nerves.

The ultrasound (US) guided erector spina plane block (ESPB) is a novel interfacial plan block defined by Forero et al. at 2016 The ESPB contains a local anesthetic injection into the deep fascia of erector spinae. This area is away from the pleural and neurological structures and thus minimizes the risk of complications due to injury. Visualization of sonoanatomy with US is easy, and the spread of local anesthetic agents can be easily seen under the erector spinae muscle. Thus, analgesia occurs in several dermatomes with cephalad-caudad way. Cadaveric studies have shown that the injection spreads to the ventral and dorsal roots of the spinal nerves. ESPB provides thoracic analgesia at the T5 level, abdominal analgesia at the T7-9 level, and lumbar analgesia at T10-12, L3 level. In the literature, it has been reported that ESPB provides effective analgesia after lumbar spine surgery.

This study aims to compare US-guided posterior QLB block and ESPB for postoperative analgesia management after lumbar disc herniation-laminectomy surgery. The primary aim is to compare postoperative pain scores (NRS) the secondary aim is to evaluate postoperative opioid consumption, motor block, and adverse effects related to opioids (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for lumbar disc herniation-laminectomy surgery under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who do not accept the procedure
* Change in surgical technique in the intraoperative period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores (NRS-Numerical Rating Scala) | Postoperative 2 hours period
  Difference in the NRS scores at postoperative 2 hours between the groups

SECONDARY OUTCOMES:
The use of rescue analgesia (number of participants) (frequency of rescue analgesia) | Postoperative 24 hours period
  Tramadol using
The use of rescue analgesia (rate of tramadol using) (total consumption) | Postoperative 24 hours period
  Tramadol using
Postoperative pain scores (NRS-Numerical Rating Scala) | Changes from baseline pain scores at postoperative 1, 4, 8, 16 and 24 hours
  The secondary aim is to compare NRS at the postoperative 1, 4, 8, 16, and 24 hours. Postoperative pain assessment will be performed using the NRS (0 = no pain, 10 = the most severe pain felt). The NRS scores will be recorded.
The incidence of adverse events | Postoperative 24 hours period
  The secondary aim is to compare the adverse events (nausea, vomiting, itching, and motor block) related to opioid agents and blocks.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Oh SK, Lim BG, Won YJ, Lee DK, Kim SS. Analgesic efficacy of erector spinae plane block in lumbar spine surgery: A systematic review and meta-analysis. J Clin Anesth. 2022 Jun;78:110647. doi: 10.1016/j.jclinane.2022.110647. Epub 2022 Jan 11. PMID 35030493
- [Background] Qiu Y, Zhang TJ, Hua Z. Erector Spinae Plane Block for Lumbar Spinal Surgery: A Systematic Review. J Pain Res. 2020 Jul 1;13:1611-1619. doi: 10.2147/JPR.S256205. eCollection 2020. PMID 32669870
- [Background] Tulgar S, Aydin ME, Ahiskalioglu A, De Cassai A, Gurkan Y. Anesthetic Techniques: Focus on Lumbar Erector Spinae Plane Block. Local Reg Anesth. 2020 Sep 25;13:121-133. doi: 10.2147/LRA.S233274. eCollection 2020. PMID 33061562
- [Background] Canikli Adiguzel S, Akyurt D, Bahadir Altun H, Ultan Ozgen G, Akdeniz S, Bayraktar B, Tulgar S, Yigit Y. Posterior Quadratus Lumborum Block or Thoracolumbar Interfascial Plane Block and Postoperative Analgesia after Spinal Surgery: A Randomized Controlled Trial. J Clin Med. 2023 Nov 21;12(23):7217. doi: 10.3390/jcm12237217. PMID 38068268
- [Background] Alver S, Ciftci B, Celik EC, Sargolzaeimoghaddam M, Cetinkal A, Erdogan C, Ahiskalioglu A. Postoperative recovery scores and pain management: a comparison of modified thoracolumbar interfascial plane block and quadratus lumborum block for lumbar disc herniation. Eur Spine J. 2024 Jan;33(1):118-125. doi: 10.1007/s00586-023-07812-3. Epub 2023 Jun 14. PMID 37314577